CLINICAL TRIAL: NCT00795249
Title: Effects of Chronic Smoking on Circulating Endothelial and Platelet-derived Microparticle
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kurume University (Other)
Responsible Party: Tsutomu Imaizumi/Chair of Cardio-vascular Medicine Kurume University, Cardio-vascular Medicine Kurume University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KurumeU-08061
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-05

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- smoker (Experimental): Individuals who have a habit of chronic smoking without any coronary risk factors
  Interventions: Behavioral: smoking cessation
- non-smoker (No Intervention): the age-matched healthy volunteers

INTERVENTIONS:
Behavioral: smoking cessation — After baseline examination, the group is asked to quit smoking for 2 weeks.
  Arms: smoker

SUMMARY:
The investigators hypothesized that circulating EMP is a useful surrogate marker of early stage of endothelial damage. To determine the effects of chronic smoking on circulating EMP, from healthy volunteers who have habit of chronic smoking, peripheral blood is drawn at the time of flow-mediated dilatation (FMD) examination. Spot urine is also collected. Circulating EMPs are counted using flow-cytometry. After 2-week smoking cessation, the measurements were repeated.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals who have no coronary risk factors

Exclusion Criteria:

* hypertension
* dyslipidemia
* chronic kidney disease
* liver dysfunction
* obesity (BMI>25.0)
* cerebrovascular disease
* other severe systemic diseases (cancer, inflammatory diseases, etc)

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The number of circulating EMP | 2 weeks

SECONDARY OUTCOMES:
FMD | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Imaizumi, MD, PhD, Study Chair — Kurume University
Locations (1):
- Kurume University Hospital, Kurume, Fukuoka, Japan